CLINICAL TRIAL: NCT06611982
Title: Guaranteed Income and Financial Treatment Trial
Brief Title: Guaranteed Income and Financial Treatment
Acronym: GIFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meredith Doherty, PhD, LCSW (Other)
Collaborators: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor-Investigator, Meredith Doherty, PhD, LCSW, Assistant Professor, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC # 31921
Record Dates: First submitted 2024-04-17; First posted 2024-09-25 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cancer; Financial Hardship; Quality of Life
MeSH Terms: conditions — Neoplasms; Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Participants assigned to the intervention arm receive $1000/month for 12 months
  Interventions: Other: Unconditional cash transfer
- Control arm (Other): Participants assigned to the control arm receive information on financial toxicity and the contact information for their social workers and financial counselors
  Interventions: Other: Contact information for social worker and financial counselor

INTERVENTIONS:
Other: Unconditional cash transfer — $1000/month for 12 months
  Arms: Intervention arm
Other: Contact information for social worker and financial counselor — Information on financial toxicity and contact information for social worker and financial counselor
  Arms: Control arm

SUMMARY:
The goal of this clinical trial is to learn if providing advanced cancer patients with $1000/month for 12 months will improve cancer outcomes. The main questions it aims to answer are:

To what extent does receiving $1000/month additional income reduce financial hardship? To what extent does receiving $1000/month additional income improve quality of life? Does receiving $1000/month additional income improve survival outcomes?

Participants will:

Receive $1000/month for 12 months Complete a survey every 3 months for 12 months If selected, participate in semi-structured interviews about their financial behaviors

DETAILED DESCRIPTION:
Cancer-related financial hardship (i.e., financial toxicity) has been associated with anxiety and depression, greater pain and symptom burden, treatment nonadherence, and mortality. Out-of-pocket healthcare costs and lost income are primary drivers of financial toxicity, however, income loss is a pronounced risk factor for cancer patients with low incomes. There has been little progress in developing an income intervention to alleviate financial toxicity cancer patients with low incomes. Unconditional cash transfers (UCT), or guaranteed income, have produced positive health effects in experiments with general low-income populations, but have not yet been evaluated in people with cancer. The Guaranteed Income and Financial Treatment (GIFT) Trial will use a two-arm randomized controlled trial to compare the efficacy of a 12-month UCT intervention providing $1000/month to treatment as usual on financial toxicity, health-related quality of life and treatment adherence in people with cancer who have low-incomes. The study will recruit 250 Medicaid beneficiaries with advanced cancer from two comprehensive cancer centers in Philadelphia, obtain informed consent, and randomize patients to one of two conditions: (1) $1,000/month UCT or (2) treatment as usual. Both arms will receive information on financial toxicity and the contact information for their hospital social worker or financial advocate upon enrollment. Participants will complete online surveys at baseline, 3, 6, 9, and 12 months from enrollment to collect patient-reported data on primary (i.e., financial toxicity, health-related quality of life, and treatment adherence) and secondary outcomes (i.e., anxiety, depression, food insecurity, housing stability). Social security records will be used to explore the effect on mortality at 2, 3, and 5 years post-enrollment. Linear mixed-models will be used to analyze all primary and secondary continuous outcomes over time and general estimating equations with a logit link and binary distribution for all binary outcomes over time. Differences between treatment and control groups and treatment effects will be determined using models that control for age, gender, race, baseline food security, baseline housing stability, and baseline ECOG. Findings from this study will have significant implications for the development and implementation of programs and policies that address the financial burden of cancer and other serious illnesses.

ELIGIBILITY:
Inclusion Criteria:

1. Age = 18 or older
2. Newly diagnosed or recurrent advanced cancer (Stage 3 or 4)
3. Receiving chemotherapy or immunotherapy (with or without radiation) at one of the recruitment sites
4. Within 12 months of receiving systemic therapy and on surveillance at one of the recruitment sites
5. ECOG performance status of 1 - 2
6. A Pennsylvania Medicaid beneficiary
7. A Pennsylvania resident

Exclusion Criteria:

1. Eligible for hospice (i.e. determined by provider to have a prognosis of 6 months or less) at time of randomization
2. Unable to communicate in English, Spanish, or Mandarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Financial Toxicity | 6 and 12 months from enrollment
  COmprehensive Score for Financial Toxicity (COST)
Treatment adherence | 6 and 12 months from enrollment
  Number of missed appointments in last 30 days

SECONDARY OUTCOMES:
Health-related quality of life | 6 and 12 months from enrollment
  Short Form Health Survey (SF-36)
Anxiety and Depression | 6 and 12 months from enrollment
  HADS
Health-related quality of life | 6 and 12 months from enrollment
  The Functional Assessment of Cancer Therapy (FACT-G)

OTHER OUTCOMES:
Mortality | 2, 3, and 5 years from enrollment
  survival time from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Doherty, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Pennsylvania Hospital, Philadelphia, New York
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Jefferson Health, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No